CLINICAL TRIAL: NCT02083523
Title: PROJECT CHOICE: Efficacy Testing of Motivational Interviewing (MI) for Adolescents Referred for Substance Use Concerns
Brief Title: Project CHOICE: Efficacy Testing of CHOICE and CHOICE+Normative Feedback Interventions
Acronym: CHOICE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Douglas Smith, Assistant Professor Douglas Smith, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Smith13356
Record Dates: First submitted 2014-01-09; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Substance-related Disorders
Keywords: Motivational Interview, normative feedback, adolescents
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interview (Active Comparator): The Motivational Interview, or MI, (15-30 minutes) was provided after initial substance use disorder assessments but prior to treatment admission. I twas facilitated by a computer generated report and included: an orientation to the session, discussion of the participants' strengths, an agenda setting procedure, a review of concerns, and a session summary. Therapists conveyed empathy, used reflective listening, tried to elicit and reinforce change talk elements, and elicited action steps from the participants.
  Interventions: Behavioral: Motivational Interview
- MI with Normative Feedback (Active Comparator): The Motivational Interview with Normative Feedback, or MI + NF, condition/intervention included all procedures described for the MI condition. Additionally, in the MI + NF condition/intervention, the participants' days of marijuana and alcohol use were compared to two sets of norms ( age specific or level of care specific) available for treatment attending youth. Therapists used whichever norm provided a greater contrast with participants' use.
  Interventions: Behavioral: Motivational Interview with Normative Feedback

INTERVENTIONS:
Behavioral: Motivational Interview with Normative Feedback — NOrmative Feedback (NF) contrasts and individual's substance use to available norms for one's reference group (i.e., descriptive norms.) Essentially, NF highlights how an individual's behavior is non-normative, which in turn, is thought to lead to reduced substance use.
  Other Names: CHOICE + (MI + NF)
  Arms: MI with Normative Feedback
Behavioral: Motivational Interview — The Motivational Interview (MI) addresses ambivalence about change. It's effects are mediated by how well counselors evoke change talk, or in-session client utterances about the: need for; commitment to; ability to; or steps needed, to change.
  Other Names: CHOICE
  Arms: Motivational Interview

SUMMARY:
This study will use a pilot test format to examine the efficacy of a brief Motivational Interviewing (MI) intervention developed by the investigator Dr. Douglas Smith called CHOICE (Compassionate Helpers Openly Inviting Client Empowerment)with youth referred for substance abuse assessments to substance abuse treatment agencies in Chicago and Urbana, IL.

DETAILED DESCRIPTION:
This study will use a pilot test format to examine the efficacy of a brief Motivational Interviewing (MI) intervention developed by the investigator Dr. Douglas Smith called CHOICE (Compassionate Helpers Openly Inviting Client Empowerment)with youth referred for substance abuse assessments to substance abuse treatment agencies in Chicago and Urbana, IL. The study will have two arms: one group will receive the standard CHOICE Motivational Interview (MI) while the second group will receive the CHOICE Motivational Interview with a Normative Feedback component, called CHOICE+ (CHOICE Plus). The hypothesis is that there will be no difference in outcomes between those that receive the standard CHOICE and those that receive the CHOICE+ MI.

ELIGIBILITY:
Inclusion Criteria:

* Youth 13-19 years of age (and their parents or legal guardians if their youth has been referred for an assessment with the Prairie Center counseling staff.)
* referred for an assessment to see if they need substance use disorder treatment
* have used substances on 13 or more days out of the past 90 days or scored higher than 2 on the CRAFT assessment. -

Exclusion Criteria:

* Low cognitive functioning

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
% Readiness to Change | Day One
  % Readiness to Change was measured immediately following receipt of the intervention session.

SECONDARY OUTCOMES:
Days of Substance Use Treatment | 3 months post intake

OTHER OUTCOMES:
Substance Use Frequency | 3 months post intake

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Smith, PhD, Principal Investigator — University of Illinois Urbana Champaign